CLINICAL TRIAL: NCT06597630
Title: Pathological Type，Gene Mutation and Clinical Characteristics of Unilateral Primary Aldosteronism，A Prospective Study
Brief Title: Pathological Type，Gene Mutation and Clinical Characteristics of Unilateral Primary Aldosteronism
Status: Recruiting | Type: Observational
Sponsor: Qifu Li (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: PGC-UPA-2024
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Aldosteronism
Keywords: Pathological type; Gene mutation
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adrenal nodule tissue specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unilateral primary aldosteronism group: The patient was diagnosed with unilateral primary aldosteronism and underwent total adrenal resection
  Interventions: Other: Tissue specimens were stained by histopathology of hematoxylin-eosin

INTERVENTIONS:
Other: Tissue specimens were stained by histopathology of hematoxylin-eosin — Whole slide images were created by scanning the complete histologic slide to produce high-resolution digital files of the histopathology of hematoxylin-eosin and CYP11B2 immunostained sections.Tissue sections of all blocks from each resected adrenal were evaluated by hematoxylin and eosin and CYP11B2 immunostaining and adrenal specimens were categorized as classical or nonclassical histopathologic findings of unilateral PA according to the HISTALDO consensus; Genotyping was performed using CYP11B2 (aldosterone synthase)-guided sequencing
  Other Names: Tissue specimens were stained by CYP11B2

SUMMARY:
1. Aim to investigate the pathological feature of UPA in Asians
2. To clarify the relationship between pathology, clinical phenotype, genetic mutation and surgical outcome of UPA in Asians.
3. To explore a new pathological type of unilateral primary aldosterone

DETAILED DESCRIPTION:
The multi-center expert team led by Tracy Ann Williams formulated the International Consensus on the Pathological Diagnosis of Unilateral aldehyde disease, which standardized the pathological classification of unilateral PA. The previous retrospective study of the research group found that the pathologic types of unilateral primary aldosteronoma were mainly classical, and aldosteronoma was the most common. There was no significant difference in clinical features and postoperative biochemical remission rate between patients with classic and non-classic, but the clinical prognosis of the latter group was worse than that of the classical group. However, the study was retrospective and there may be inclusion bias. The pathologic distribution and clinical features of unilateral aldehyde disease are not completely clear and need to be discussed in prospective studies.Therefore，this study aims to determine the composition ratio of different pathological types in patients with unilateral procaldosis enrolled in our center. Gene mutation of different pathological types, the relationship between pathology and clinical phenotype, gene mutation, etc.

ELIGIBILITY:
Inclusion Criteria:

1. No gender limitation;
2. Age 18-80 years old;
3. The patient was diagnosed with UPA and underwent total adrenal resection.

Exclusion Criteria:

1. Bilateral disease
2. Partial of no biochemical response in follow-up
3. partial adrenalectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, about 100 patients with unilateral protonaldehydes undergoing total adrenal resection will be continuously enrolled in this research center from December 2023.
  Unilateral Primary Aldosteronism underwent total Adrenalectomy were continuously included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Define the aldosterone-producing adenoma and aldosterone-producing nodule(classical)proportions | 2 weeks after surgery
  Adrenal operative specimens were diagnosed as aldosterone-producing adenoma、aldosterone-producing nodule、aldosterone-producing micronodules、aldosterone-producing diffusehyperplasia according to HE and CYP11B2 staining
The proportion with genetic mutations | 2 weeks after surgery
  The adrenal tumor was diagnosed by gene sequencing as KCNJ5 mutation, ATP1A1 mutation, ATP2B3 mutation or CACNA1D mutation,etc.
Analyze the Aldosterone level and renin level Characteristics | 2 weeks after surgery
  Aldosterone level（pg/ml）, renin level（uIU/ml）, blood potassium（mmol/L） and blood pressure are the main clinical indicators of primary aldosteronism(Aldosterone level divided by renin level to obtain ARR, ARR greater than 20 consider whether aldosterone autonomic secretion),different pathological types of aldosteronomas were measured to analyze whether there were differences in clinical characteristics of adrenal tumors of different pathological types

SECONDARY OUTCOMES:
Define the ldosterone-producing micronodules and aldosterone-producing diffusehyperplasia(Nonclassical)proportions | 2 weeks after surgery
  Adrenal operative specimens were diagnosed as aldosterone-producing adenoma、aldosterone-producing nodule、aldosterone-producing micronodules、aldosterone-producing diffusehyperplasia according to HE and CYP11B2 staining
Analyze the blood potassium and blood pressure Characteristics | 2 weeks after surgery
  Primary aldosterone has varying degrees of hypertension with or without hypokalemia

CONTACTS AND LOCATIONS:
Overall Officials: Li Qifu, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Qifu Li, PhD, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi GP, Sechi LA, Giacchetti G, Ronconi V, Strazzullo P, Funder JW. Primary aldosteronism: cardiovascular, renal and metabolic implications. Trends Endocrinol Metab. 2008 Apr;19(3):88-90. doi: 10.1016/j.tem.2008.01.006. Epub 2008 Mar 7. PMID 18314347
- [Background] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Background] Yang Y, Xiao M, Song Y, Tang Y, Luo T, Yang S, He W, Cheng Q, Ma L, Zhang Y, He Y, Cao Y, Yang J, Peng B, Hu J, Li Q. H-score of 11beta-hydroxylase and aldosterone synthase in the histopathological diagnosis of adrenocortical tumors. Endocrine. 2019 Sep;65(3):683-691. doi: 10.1007/s12020-019-02022-8. Epub 2019 Jul 22. PMID 31332713
- [Background] Yamazaki Y, Omata K, Tezuka Y, Ono Y, Morimoto R, Adachi Y, Ise K, Nakamura Y, Gomez-Sanchez CE, Shibahara Y, Kitamoto T, Nishikawa T, Ito S, Satoh F, Sasano H. Tumor Cell Subtypes Based on the Intracellular Hormonal Activity in KCNJ5-Mutated Aldosterone-Producing Adenoma. Hypertension. 2018 Sep;72(3):632-640. doi: 10.1161/HYPERTENSIONAHA.118.10907. PMID 30354756
- [Background] Sun N, Meyer LS, Feuchtinger A, Kunzke T, Knosel T, Reincke M, Walch A, Williams TA. Mass Spectrometry Imaging Establishes 2 Distinct Metabolic Phenotypes of Aldosterone-Producing Cell Clusters in Primary Aldosteronism. Hypertension. 2020 Mar;75(3):634-644. doi: 10.1161/HYPERTENSIONAHA.119.14041. Epub 2020 Jan 20. PMID 31957522
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Result] Funder JW. Primary aldosteronism as a public health issue. Lancet Diabetes Endocrinol. 2016 Dec;4(12):972-973. doi: 10.1016/S2213-8587(16)30272-8. No abstract available. PMID 27886747
- [Result] Mete O, Asa SL, Giordano TJ, Papotti M, Sasano H, Volante M. Immunohistochemical Biomarkers of Adrenal Cortical Neoplasms. Endocr Pathol. 2018 Jun;29(2):137-149. doi: 10.1007/s12022-018-9525-8. PMID 29542002
- [Result] Nishimoto K, Koga M, Seki T, Oki K, Gomez-Sanchez EP, Gomez-Sanchez CE, Naruse M, Sakaguchi T, Morita S, Kosaka T, Oya M, Ogishima T, Yasuda M, Suematsu M, Kabe Y, Omura M, Nishikawa T, Mukai K. Immunohistochemistry of aldosterone synthase leads the way to the pathogenesis of primary aldosteronism. Mol Cell Endocrinol. 2017 Feb 5;441:124-133. doi: 10.1016/j.mce.2016.10.014. Epub 2016 Oct 14. PMID 27751767
- [Result] Gomez-Sanchez CE, Kuppusamy M, Reincke M, Williams TA. Disordered CYP11B2 Expression in Primary Aldosteronism. Horm Metab Res. 2017 Dec;49(12):957-962. doi: 10.1055/s-0043-122238. Epub 2017 Dec 4. PMID 29202495
- [Result] Nishimoto K, Nakagawa K, Li D, Kosaka T, Oya M, Mikami S, Shibata H, Itoh H, Mitani F, Yamazaki T, Ogishima T, Suematsu M, Mukai K. Adrenocortical zonation in humans under normal and pathological conditions. J Clin Endocrinol Metab. 2010 May;95(5):2296-305. doi: 10.1210/jc.2009-2010. Epub 2010 Mar 3. PMID 20200334
- [Result] Williams TA, Gomez-Sanchez CE, Rainey WE, Giordano TJ, Lam AK, Marker A, Mete O, Yamazaki Y, Zerbini MCN, Beuschlein F, Satoh F, Burrello J, Schneider H, Lenders JWM, Mulatero P, Castellano I, Knosel T, Papotti M, Saeger W, Sasano H, Reincke M. International Histopathology Consensus for Unilateral Primary Aldosteronism. J Clin Endocrinol Metab. 2021 Jan 1;106(1):42-54. doi: 10.1210/clinem/dgaa484. PMID 32717746
- [Result] Monticone S, Castellano I, Versace K, Lucatello B, Veglio F, Gomez-Sanchez CE, Williams TA, Mulatero P. Immunohistochemical, genetic and clinical characterization of sporadic aldosterone-producing adenomas. Mol Cell Endocrinol. 2015 Aug 15;411:146-54. doi: 10.1016/j.mce.2015.04.022. Epub 2015 May 6. PMID 25958045
- [Result] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687